CLINICAL TRIAL: NCT00754689
Title: A Multicenter, Double Blind, Placebo Controlled Randomized Study of the Efficacy and Safety of Two Rimonabant/Metformin Combinations for Reducing A1C in the Treatment of Patients With Type 2 Diabetes Mellitus Who Are Not on Current Drug Therapy.
Brief Title: Study of Rimonabant/Metformin Combinations to Investigate Diabetes (Blood Sugar) Control in Patients With Type 2 Diabetes
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision taken in light of demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC10231; 2008-002500-26 (EudraCT Number)
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Rimonabant/metformin combination
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rimonabant; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1 (Active Comparator): Metformin 500mg twice daily (bid) + placebo
  Interventions: Drug: Metformin; Drug: placebo
- Arm 2 (Active Comparator): Metformin 1000mg bid + placebo
  Interventions: Drug: Metformin; Drug: placebo
- Arm 3 (Active Comparator): Rimonabant 20mg once daily (od) + placebo
  Interventions: Drug: Rimonabant; Drug: placebo
- Arm 4 (Experimental): Rimonabant 10mg bid (from week 2) in combination with metformin 500mg bid
  Interventions: Drug: Rimonabant; Drug: Metformin
- Arm 5 (Experimental): Rimonabant 10mg bid (from week 2) in combination with metformin 1000mg bid
  Interventions: Drug: Rimonabant; Drug: Metformin

INTERVENTIONS:
Drug: Rimonabant — Tablet, oral administration
  Other Names: SR141716; Acomplia
  Arms: Arm 3; Arm 4; Arm 5
Drug: Metformin — Tablet, oral administration
  Arms: Arm 1; Arm 2; Arm 4; Arm 5
Drug: placebo — Tablet, oral administration
  Arms: Arm 1; Arm 2; Arm 3

SUMMARY:
The primary objective of the study is to demonstrate superiority of rimonabant/metformin combinations in Glycosylated Hemoglobin 1c (A1C) reduction over the corresponding single agent metformin and over rimonabant alone in patients with type 2 diabetes mellitus at 9 months.

The secondary objective is to investigate the effects of rimonabant/metformin combinations for reducing fasted plasma glucose, body weight and triglycerides, and raising High Density Lipoprotein Cholesterol (HDL-C) in comparison with metformin at 9 months.

Another objective is to evaluate the safety of rimonabant in combination with metformin over a period of up to 52 weeks.

DETAILED DESCRIPTION:
The duration per patient is up to 65 weeks: 1 - 2 weeks screening, up to 52 weeks double blind treatment, and 75 days post last dose. This study will end for all patients when the last patient has been treated for at least 9 months.

ELIGIBILITY:
Inclusion Criteria:

* History of type 2 diabetes mellitus diagnosed prior to the screening visit 1 (ADA criteria)
* Patients must not have used any oral or injectable glucose lowering medication at least 12 weeks prior to the screening visit to establish a stable, comparable baseline A1C assessment in all patients
* A1C ≥7.0 % and ≤10.0 %
* Fasted plasma glucose at screening visit ≤260 mg/dL (14.44 mmol/L)

Exclusion Criteria:

* Treatment with any anti-diabetic oral agent, or injectable antidiabetic agent within 12 weeks prior to screening visit
* In the 3 months prior to the screening visit, use of any anti-obesity agent or drugs for weight loss, or administration of systemic corticosteroids for more than 7 days
* Presence of any severe medical or psychological condition that, in the opinion of the investigator, would compromise the patient's safe participation including uncontrolled serious psychiatric illness such a major depression within the last 2 years, and history of other severe psychiatric disorders
* Presence or history of cancer within the past five years
* Pregnant or breast-feeding women, or women of childbearing potential not protected by effective method of birth control

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in A1C | at 9 months

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose | at 9 months
Change from baseline in body weight | at 9 months
Percent change from baseline in triglycerides | at 9 months
Percent change from baseline in HDL-C | at 9 months

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States